CLINICAL TRIAL: NCT02002130
Title: The Use of Glutamic Acid Decarboxylase (GAD)and Gamma-Amino Butyric Acid(GABA)in the Treatment of Type I Diabetes.
Brief Title: The Use of Glutamic Acid Decarboxylase (GAD) and Gamma-Amino Butyric Acid (GABA) in the Treatment of Type I Diabetes
Acronym: GABA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Diamyd Inc (Industry); NOW Foods (Other); Janssen Pharmaceuticals (Industry); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Kenneth McCormick, MD, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GABA-GAD
Record Dates: First submitted 2013-11-18; First posted 2013-12-05 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Type I Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo GABA and Placebo GAD-alum (Placebo Comparator): Placebo formulation, Maltodextrin, for Gamma-Amino Butyric Acid (GABA) capsule-identical in appearance and taste, but no active medication will be taken with meals.Number of pills based on body surface area.
  Placebo GAD-alum(Glutamic Acid Decarboxylase in alum) injection- identical in appearance but no active medication will be received at baseline and 1 month.
  Interventions: Drug: Placebo GABA and Placebo GAD-alum
- GABA and placebo GAD-alum (Active Comparator): Patients will receive the Active GABA (Gamma-Amino Butyric Acid) capsules. Each capsule 250mg. Dosage will be calculated according to body surface area of the child and divided between 2 meals/day. Larger dose taken with larger meal.
  Patients will receive the GAD-alum( Glutamic Acid Decarboxylase in alum) placebo at baseline and 1 month.
  Interventions: Drug: GABA and Placebo GAD-alum
- Active Oral GABA and Active GAD-alum Injection (Active Comparator): Patients will receive Oral GABA(Gamma-Amino Butyric Acid) 250mg capsules. Dosage (# of capsules) based on body surface area and divided between 2 meals/day.
  Patients will receive a primary (at baseline)injection of recombinant human GAD(Glutamic Acid Decarboxylase) in a standard vaccine formulation with alum, and a booster injection of the same at 1 month after baseline.
  Interventions: Drug: Active Oral GABA and Active GAD-alum injection

INTERVENTIONS:
Drug: Placebo GABA and Placebo GAD-alum — Maltodextrin as a placebo formulation for GABA Placebo GAD-alum injection
  Other Names: Placebo for Gamma-Amino Butyric Acid
  Arms: Placebo GABA and Placebo GAD-alum
Drug: GABA and Placebo GAD-alum — Oral Active GABA with Placebo GAD-alum
  Arms: GABA and placebo GAD-alum
Drug: Active Oral GABA and Active GAD-alum injection — Active Oral GABA and Active GAD-alum injection
  Arms: Active Oral GABA and Active GAD-alum Injection

SUMMARY:
Type I Diabetes is an auto immune disease in which the body's immune system attacks and destroys the insulin-producing beta cells of the pancreas. Therefore, children affected by this condition present with high blood sugars. This condition affects 1:400/500 persons worldwide.Type I Diabetes, previously known as Juvenile Diabetes,usually strikes in childhood, adolescence, or young adulthood, but lasts for a lifetime. To date, there has been no treatments that can arrest, or reverse the ongoing beta cell destruction. We hypothesize that GABA, a naturally occurring substance, has the potential to reduce the inflammation and protect the pancreatic beta cells from autoimmune destruction. GAD-alum may contribute to the preservation of residual insulin secretion in patients with recent onset, Type I Diabetes.

DETAILED DESCRIPTION:
The primary defect in autoimmune Type I Diabetes Mellitus (T1DM) involves the infiltration of the pancreatic islet cells by T-lymphocytes, macrophages, and other immune cells, and consequent loss of beta cells. At the onset of T1DM more than 70% of the beta cells are destroyed, whereas the residual beta cells most likely represent the only reservoir for the potential regeneration of the islet beta cell mass. A series of immunological abnormalities have been reported in those with T1DM including, but not limited to, the production of autoantibodies (i.e., glutamic acid decarboxylase (GAD-65), tyrosine phosphatase-related islet antigen 2 (IA2), Zinc Transporter 8 (ZnT8A), or insulin (IAA) as well as alterations in the capacity of regulatory T cells (Treg) to suppress the action of effector T cells (Teff); the latter population thought as playing a key role in the immune destructive process. Therefore, a vast majority of studies attempting to prevent or reverse the disease have focused on immune suppression. While some of these studies have shown limited promise, many has side effects which were significant enough that one must question the value of short term benefits associated with utilizing these drugs.

GABA is a naturally occurring substance in physiology and has the potential to locally reduce inflammation and protect pancreatic beta cells from auto-immune destruction. GABA, synthesized from glutamate by GAD, is a well known neurotransmitter in the CNS and acts mainly through the GABAA receptor (GABAAR). GABA is locally produced by the pancreatic beta cells. GABAARs are also expressed in various immune cells, including T-cells, peripheral blood mononuclear cells, and are known to exert immune-inhibitory effects. BABA appears to play multiple roles in the pancreas. GABA promotes beta-cell growth and survival, and GABA can also act on the GABA(A) receptors in the pancreatic alpha cells, in so doing suppressing glucagon secretion, and GABA suppresses inflammation and increases regulatory T-cell numbers. Based on the aforementioned information, we envisage that administering GABA to those with new onset T1DM may preserve or increase residual insulin production, suppress glucagon release, and decrease inflammation surrounding the pancreas. With this, GABA may prolong the beta-cell life after diagnosis. Combining with GAD-alum injections, which aim to halt the autoimmune attack by inducing tolerance thereby saving residual insulin production, may improve glycemic control even more and significantly decrease the risk of hypoglycemia and long-term complications in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be positive for GAD-65 antibody.
* They must meet ADA criteria for diabetes: classic symptoms, plus blood sugar > 200mg/dL or fasting blood sugar > 126 mg/dL.
* Must be enrolled with 5 weeks of diagnosis
* Females who are post-menarchal must use 2 forms of contraception if not abstinent. The types of contraception deemed acceptable would be oral contraceptives, intrauterine devices, and barrier methods.
* Signed informed consent form.

Exclusion Criteria:

* Chronic systemic steroid use, including inhaled compounds, or any medication which can alter glucose metabolism
* Obesity, defined as BMI > 95% or BMI > 27 in adolescents with acanthosis score between 1-1.5.
* Pregnant and/or breast feeding
* History of seizure disorder
* Patients on medications that may disturb GABA action, such as Baclofen, Valium, Acamprosate, Neurontin, or Lyrica
* history of any alcoholism or substance abuse.
* Chronic Disease (such as liver, cancer, cystic fibrosis, or renal failure)
* Chromosome abnormality (such as Trisomy 21, Turner Syndrome, etc.)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Compare the effect of oral GABA or oral GABA/GAD combination administration on pancreatic beta cell function by quantitative C-peptide secretion | 12 months after baseline
  This will be assessed by meal stimulated c-peptide secretion in treatment cohorts compared to age matched placebo controls before and after 1 year of treatment.

SECONDARY OUTCOMES:
Compare the effect of oral GABA or GABA/GAD administration on fasting and meal stimulated glucagon and pro-insulin levels. | 12 months after baseline
  This will be assessed by meal stimulated glucagon and pro-insulin secretion in treatment cohorts compared with age matched placebo controls before and after 1 year of treatment.
Compare the effect of oral GABA or GABA/GAD administration on total daily insulin usage by participants and corrected Hemoglobin A1C. | 12 months after baseline
  This will be assessed by measuring insulin usage and corrected Hemoglobin A1C linearly for each participant, in addition to comparison with age matched controls
Compare the effect of oral GABA or oral GABA/GAD administration on indices of immune system function. | 12 months after baseline
  This will be assessed by measuring immunologic markers of inflammation linearly over the 12 month treatment course for each patient and comparing to age matched placebo controls.
Compare the effect of oral GABA or oral GABA/GAD administration on diabetes related autoantibodies | 12 months after baseline
  This will be assessed by measuring GAD65, ICA512, and Zinc Transporter 8 antibodies throughout the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth McCormick, MD, Principal Investigator — University of Alabama at Birmingham; Gail Mick, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Background] Ludvigsson J, Faresjo M, Hjorth M, Axelsson S, Cheramy M, Pihl M, Vaarala O, Forsander G, Ivarsson S, Johansson C, Lindh A, Nilsson NO, Aman J, Ortqvist E, Zerhouni P, Casas R. GAD treatment and insulin secretion in recent-onset type 1 diabetes. N Engl J Med. 2008 Oct 30;359(18):1909-20. doi: 10.1056/NEJMoa0804328. Epub 2008 Oct 8. PMID 18843118
- [Background] Soltani N, Qiu H, Aleksic M, Glinka Y, Zhao F, Liu R, Li Y, Zhang N, Chakrabarti R, Ng T, Jin T, Zhang H, Lu WY, Feng ZP, Prud'homme GJ, Wang Q. GABA exerts protective and regenerative effects on islet beta cells and reverses diabetes. Proc Natl Acad Sci U S A. 2011 Jul 12;108(28):11692-7. doi: 10.1073/pnas.1102715108. Epub 2011 Jun 27. PMID 21709230
- [Derived] Heath KE, Feduska JM, Taylor JP, Houp JA, Botta D, Lund FE, Mick GJ, McGwin G Jr, McCormick KL, Tse HM. GABA and Combined GABA with GAD65-Alum Treatment Alters Th1 Cytokine Responses of PBMCs from Children with Recent-Onset Type 1 Diabetes. Biomedicines. 2023 Jul 10;11(7):1948. doi: 10.3390/biomedicines11071948. PMID 37509587
- [Derived] Freese J, Al-Rawi R, Choat H, Martin A, Lunsford A, Tse H, Mick G, McCormick K. Proinsulin to C-Peptide Ratio in the First Year After Diagnosis of Type 1 Diabetes. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4318-e4326. doi: 10.1210/clinem/dgab463. PMID 34228132

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT02002130/Prot_SAP_000.pdf